CLINICAL TRIAL: NCT02678598
Title: A Retrospective Study Evaluating the Efficacy and Safety of Micafungin Sodium in the Treatment of Invasive Fungal Infections
Status: Completed | Type: Observational
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9463-MA-3003
Record Dates: First submitted 2016-02-02; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Invasive Fungal Infections
Keywords: Micafungin; Candida; Aspergillosis; Antifungal
MeSH Terms: conditions — Invasive Fungal Infections; Torulopsis; Aspergillosis | interventions — Micafungin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Micafungin group
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Intravenous

SUMMARY:
The objective of this study is to evaluate the efficacy of intravenous micafungin for the empirical antifungal therapy, pre-emptive antifungal therapy, diagnostic driven antifungal therapy or targeted antifungal therapy patients with invasive fungal infections caused by Candida sp. or Aspergillus sp. (fungemia, respiratory mycosis, gastrointestinal mycosis) in adult patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Micafungin as empirical antifungal therapy, pre-emptive antifungal therapy, diagnostic driven antifungal therapy or targeted antifungal therapy
* Patients received Micafungin treatment at least 1 dose

Exclusion Criteria:

* Patients received Micafungin treatment combined with other antifungal drugs at the same time
* Neither efficacy or safety can be evaluated because of missing data, confused record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The hospitalized patients who received intravenous micafungin for treatment according to the clinical judgment of the treating physician before the end of April 2015
Sampling Method: Non-Probability Sample
Enrollment: 2555 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall success rate | Up to 12 months
  Overall success rate=number of overall success patients/number of patients for efficacy evaluation × 100%

SECONDARY OUTCOMES:
Overall incidence and severity of adverse events | Up to 12 months
Overall incidence and severity of adverse drug reactions | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma China, Inc.
Locations (17):
- China (17):
  - Beijing
  - Changchun
  - Chengdu
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Guizhou
  - Haikou
  - Hangzhou
  - Harbin
  - Hengyang
  - Langfang
  - Shanghai
  - Shijiazhuang
  - Wuhan
  - Xiamen
  - Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng X, Huang X, Luo J, Li J, Li W, Liu Q, Niu T, Wang X, Zhou J, Zhang X, Hu J, Liu K. Effectiveness and Tolerability of Micafungin in Chinese Patients with Invasive Fungal Infections: A Retrospective, Multicenter Study. Adv Ther. 2018 Sep;35(9):1400-1410. doi: 10.1007/s12325-018-0762-5. Epub 2018 Aug 13. PMID 30105657